CLINICAL TRIAL: NCT02730754
Title: Relationship Between Emotional Disorders (Diabetes Distress and Depression) and Outcomes (Self-care and Clinical) in Adults With Type 2 Diabetes Mellitus in Primary Care: A Retrospective Cohort Study
Brief Title: Emotional Disorders and Outcomes in Adults With Type 2 Diabetes Mellitus at Primary Care
Acronym: EDDMQoL-Pro
Status: Completed | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Boon-How Chew, Associate Professor, Universiti Putra Malaysia
Other Study IDs: NMRR-15-2214-28139
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Mood Disorders; Illness Perception; Primary Care; Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Mood Disorders; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to determine which factors are related to change in diabetes-related distress and change in depressive symptoms after three years of follow-up in Asian adults with type 2 diabetes mellitus in primary care. The investigators will explore the impact of patient demographics, cardiometabolic control, medications adherence, health-related quality of life, self-efficacy and self-management behaviors on diabetes-related distress and depressive symptoms.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus (T2DM) have been shown to experience psychological burden and distorted illness perception. These psychological burden include feeling of burned-out, fatigue, distress and depression, and in addition of distorted illness perception often lead to difficulty in coping with the demands of life-style changes and adherence to medication. Diabetes-related distress (DRD) and depressive symptoms (DS) were associated with glycaemic control and medication adherence, and life-styles behaviors, respectively. However, evidence on the relationships between DRD, DS and clinically significant outcomes are scarce in Asian adults with T2DM. Primary care patients who participated before will be re-invited. This is a repeated cross-sectional study of a cohorts of 700 patients who were first studied in 2013 (Emotional Distress in adults with type 2 Diabetes Mellitus & Quality of Life [EDDMQoL] study with the National Medical Research Register (NMRR) identification number: NMRR-12-1167-14158). Demographic data (age, gender, ethnicity, religion, educational level, occupation and monthly income), smoking status, self-perceive social support and health literacy will be collected by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Those who participated in the EDDMQoL study
2. Adults aged at least 30 year-old
3. Diagnosed of T2DM more than three years ago
4. On regular follow-up with at least three visits in the previous year

Exclusion Criteria:

1. Patients who are pregnant or lactating
2. Having psychiatric/psychological disorders that could impair judgments and memory
3. Patients who cannot read or understand English, Malay or Mandarin

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated before in the EDDMQoL in 2013 (NMRR ID: NMRR-12-1167-14158)
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Diabetes-related distress measured with Diabetes Distress Scale-17 | Baseline and 3 year
  Change in diabetes-related distress
Depressive symptoms measured with Patient Health Questionnaire-9 | Baseline and 3 year
  Change in depressive symptoms

SECONDARY OUTCOMES:
Diabetes-related distress and depression combined | Baseline and 3 year
  Change in both diabetes-related distress and depressive symptoms combined
Illness perceptions measured with Brief Illness Perception Questionnaire | Through study completion
  Cross-sectional, an association with other variables
Diabetes distress measured with Problem Areas in Diabetes Scale (PAID-5) | Through study completion
  Cross-sectional, an association with other variables

OTHER OUTCOMES:
Variability in HbA1c | Baseline and 3-year
  Standard deviations of the HbA1c from the medical records
Variability in systolic blood pressure | Baseline and 3-year
  Standard deviations of the systolic blood pressures from the medical records
Variability in pulse rates | Baseline and 3-year
  Standard deviations of the pulse rates from the medical records
Health care utilisation/hospitalisation | 3-year
  Retrospective records of the number of visits to healthcare facilities and hospitalisation from the medical records

CONTACTS AND LOCATIONS:
Overall Officials: Boon How Chew, MMed, Principal Investigator — Universiti Putra Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be made available in figshare

REFERENCES:
- [Background] Chew BH, Vos RC, Stellato RK, Rutten GEHM. Diabetes-Related Distress and Depressive Symptoms Are Not Merely Negative over a 3-Year Period in Malaysian Adults with Type 2 Diabetes Mellitus Receiving Regular Primary Diabetes Care. Front Psychol. 2017 Oct 17;8:1834. doi: 10.3389/fpsyg.2017.01834. eCollection 2017. PMID 29089913
- [Background] Chew BH, Vos RC, Pouwer F, Rutten GEHM. The associations between diabetes distress and self-efficacy, medication adherence, self-care activities and disease control depend on the way diabetes distress is measured: Comparing the DDS-17, DDS-2 and the PAID-5. Diabetes Res Clin Pract. 2018 Aug;142:74-84. doi: 10.1016/j.diabres.2018.05.021. Epub 2018 May 24. PMID 29802952
- [Result] Chew BH, Vos RC, Heijmans M, Shariff-Ghazali S, Fernandez A, Rutten GEHM. Validity and reliability of a Malay version of the brief illness perception questionnaire for patients with type 2 diabetes mellitus. BMC Med Res Methodol. 2017 Aug 3;17(1):118. doi: 10.1186/s12874-017-0394-5. PMID 28774271
- [Derived] Chew BH, Hussain H, Supian ZA. Is therapeutic inertia present in hyperglycaemia, hypertension and hypercholesterolaemia management among adults with type 2 diabetes in three health clinics in Malaysia? a retrospective cohort study. BMC Fam Pract. 2021 Jun 11;22(1):111. doi: 10.1186/s12875-021-01472-2. PMID 34116645